CLINICAL TRIAL: NCT07396649
Title: Feasibility of Non-invasive Electrical Nerve Stimulation of the Upper Airway in Patients With Obstructive Sleep Apnoea
Brief Title: Feasibility of Upper Airway Stimulation in OSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Notos Medical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIV-25-10-054794; Project Breathe 1 (Other: Notos Medical Limited)
Record Dates: First submitted 2026-01-20; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Obstructive Sleep Apnoea (OSA)
Keywords: obstructive sleep apnoea; OSA; sleep apnoea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Masking Description: Assessors scoring the drug induced sleep endoscopy VOTE videos will be blinded to the treatment provided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-invasive electrical stimulation of the upper airway (Experimental): Participants will have bilateral non-invasive electrical stimulation of the submandibular region while undergoing a polysomnography assessment and during drug induced sleep endoscopy.
  Interventions: Device: Non-invasive electrical stimulation

INTERVENTIONS:
Device: Non-invasive electrical stimulation — The non-invasive electrical stimulation components will consist of two Digitimer DS5 isolated current stimulators, voltage control by an NI-9262 module, and two pairs of adhesive electrodes placed in the submandibular region.
  Other Names: Breathe Study System

SUMMARY:
Project Breathe 1 is a short-duration (5 month) pilot investigation to assess the safety and tolerability of non-invasive electrical stimulation in adults with obstructive sleep apnoea. The investigation is an unblinded, uncontrolled, single arm design.

ELIGIBILITY:
Inclusion Criteria:

* Obstructive sleep apnoea diagnosis with an AHI of 15-50 events/hour recorded in the baseline polysomnography (PSG)
* BMI < 32 kg/m²
* Age > 18 years old
* Able to read, write, and speak Dutch with acceptable visual and auditory acuity
* Able and willing to provide informed consent

Exclusion Criteria:

* Presence of a cardiac pacemaker or implantable cardiac defibrillator or ventriculoperitoneal shunt
* Central (non-obstructive) AHI episodes >5 events/hour recorded in the baseline PSG
* Inability to sleep supine
* Pregnancy
* Inability to undergo DISE
* Inability or unwillingness to shave under and around their chin and neck if appropriate
* Known inability to complete PSG with a total sleep time of > 4 hours
* The use of other neurostimulatory devices
* A diagnosis of periodic leg movement disorder
* Awake resting arterial oxygen saturation <93% (suggesting possible hypoventilation)
* Unstable, untreated coronary or peripheral artery disease
* Severe arterial hypertension defined as a resting blood pressure (BP) of >180/110mmHg
* Currently employed as a professional driver
* Any previous sleep-related driving accident
* A past or current condition that in the opinion of the investigator contraindicates enrolment (e.g. chronic substance abuse, severe psychiatric disorders)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-29 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Tolerability of non-invasive electrical stimulation of the upper airway during sleep | Night 1
  The proportion of participants who are able to tolerate 80% of their maximum awake tolerated dose during sleep.

SECONDARY OUTCOMES:
Arousals | Night 1
  Number of arousals during sleep when patient is undergoing non-invasive electrical stimulation of the upper airway during respiratory events.
Subjective awareness of stimulation during sleep | Night 1
  Number of actual stimulation events compared to number of events felt by the participant. Number of subjective events will be determined post-sleep.

OTHER OUTCOMES:
Respiratory disturbance index | Baseline, Night 1
  Number of arousals from respiratory events. Only arousals during which stimulation was initiated will be included.
Apnoea-Hypopnoea Index | Baseline, Night 1
  Number of apneas and hypopneas per hour of sleep.
Oxygen desaturation index | Baseline, Night 1
  Number of desaturations (drop in oxygen saturation >3%) per hour of sleep
Drug induced sleep endoscopy | Day 3
  The VOTE classification system defines the degree of upper airway collapse at the level of the Velum (V), Oropharynx (O), Tongue (T) and Epiglottis (E). Collapse will be defined as either complete obstruction (2), partial obstruction (1) or no obstruction (0) at each level, and the pattern of collapse will be described at each level (antero-posterior for VTE, lateral for VOE, or concentric for V). Scoring will be conducted by three Investigators blinded to treatment allocation (i.e. baseline or with electrical stimulation). The three expert Investigators will review and come to consensus on scoring for each video.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Verbraecken, Principal Investigator — Universiteit Antwerpen
Locations (1):
- Antwerp University Hospital, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No